CLINICAL TRIAL: NCT01166958
Title: Enhancing Osteoporosis Therapy: Can We Open the Anabolic Window?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-2010-0064
Record Dates: First submitted 2010-07-15; First posted 2010-07-21 (Estimated); Results first posted 2014-09-22 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Teriparatide; Raloxifene Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Daily teriparatide (Forteo) (Active Comparator)
  Interventions: Drug: Teriparatide
- Monthly cycles of teriparatide followed by raloxifene (Active Comparator)
  Interventions: Drug: Teriparatide; Drug: Raloxifene

INTERVENTIONS:
Drug: Teriparatide — Teriparatide (TPD; Forteo) is supplied as a pre-filled syringe that dispenses 20 ug. The dose is one subcutaneous injection daily. Each pre-filled injection delivery device contains sufficient TPD for a 28-day supply of 20 mcg/day.
  Other Names: Forteo
Drug: Raloxifene — Raloxifene (RLX; Evista) is supplied as a 60 mg tablet. RLX is stored at room temperature.
  Other Names: Evista
  Arms: Monthly cycles of teriparatide followed by raloxifene

SUMMARY:
Current osteoporosis therapies produce a prompt increase in bone mass, followed by only modest or no further subsequent gains. This limitation, known as the "remodeling transient," reflects the "coupling" of bone resorption with formation such that interventions impacting either of these processes lead to compensatory changes of the other. For example, medications which increase bone formation promptly also stimulate bone resorption. Thus, given the need to dramatically increase bone mass in patients with osteoporosis, it is necessary to "uncouple" formation and resorption. The investigators believe this to be possible using currently existing FDA-approved therapeutic agents, by using a novel, sequential approach.

This pilot project will obtain preliminary data essential to support future work. In this study, the investigators will begin to explore the use of sequential anabolic treatment with teriparatide followed by antiresorptive therapy with raloxifene. The investigators propose that such sequential treatment will allow opening of the "anabolic window," the brief period of time following initiation of teriparatide therapy in which bone formation exceeds resorption.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy, community-dwelling ambulatory post-menopausal women.
* Able and willing to sign informed consent.
* Age 60 to 89.
* Have osteoporosis defined as follows:
* BMD T-score of the lumbar spine, femur neck, total proximal femur or .3 radius of -2.5 to -4.0; note: the lumbar spine must include two vertebrae that are evaluable by DXA in the opinion of the investigator.

OR

* BMD T-score of the lumbar spine, femur neck, total proximal femur or .3 radius of -1.5 or lower and either an atraumatic (in the opinion of the investigator) nonvertebral fracture; [note: nonvertebral fracture sites include the wrist, hip, pelvis, ribs, humerus, clavicle, femur, tibia and fibula] or a minimum of two mild or one moderate or severe atraumatic vertebral fractures (defined using the Genant visual semi-quantitative scale).
* Baseline serum 25(OH)D concentration > 20 ng/ml and < 60 ng/ml.
* Able and willing to receive daily subcutaneous injections using a Forteo® pen.

Exclusion Criteria:

* History of exposure to external beam or implant radiation therapy involving the skeleton.
* Paget's disease or unexplained elevations of alkaline phosphatase.
* Any history of venous thrombosis including deep vein thrombosis, pulmonary embolism, retinal vein thrombosis and superficial phlebitis.
* Documented atherosclerotic vascular disease, including but not limited to prior myocardial infarction, angina, atrial fibrillation, stroke and TIA.
* Marked hypertriglyceridemia (>500 mg/dl).
* History of prior treatment with estrogen resulting in hypertriglyceridemia (> 500 mg/dl).
* Serum calcium, alkaline phosphatase, PTH or TSH outside the normal reference range.
* History of nephrolithiasis or urolithiasis within 10 years prior to enrollment; those with a history of nephro- or urolithiasis must have an appropriate radiology study (e.g., IVP or KUB) within six months documenting absence of stones.
* Baseline 24-hour urine calcium > 250 mg.
* Known risk factors for hypercalcemia, e.g., malignancy, tuberculosis, sarcoidosis.
* History of any form of cancer except adequately treated squamous cell or basal cell skin carcinoma.
* Use of active vitamin D analogs or high dose vitamin D (≥50,000 IU weekly) in the last year.
* Active or suspected diseases (within 1 year prior to enrollment) that affect bone metabolism, e.g., renal osteodystrophy, hyperthyroidism, osteomalacia, hyperparathyroidism.
* Known allergy, hypersensitivity, contraindication or intolerance to teriparatide or raloxifene.
* History of vaginal bleeding within the past year.
* Renal failure or substantial hepatic impairment. Note "renal failure" is defined as a calculated creatinine clearance (using the Cockroft-Gault formula) of ≤ 35 ml/minute.
* Severe disease, e.g., cardiac, hepatic, pulmonary, etc., which may limit ability to complete this study. Specifically, significantly impaired hepatic function (ALT or GGT 3x the upper limit of normal.
* Known malabsorption syndromes, e.g., celiac disease, active inflammatory bowel disease, gastric bypass, etc.
* Use of anion exchange resins (e.g., cholestyramine) in the past month.
* Current use of warfarin (coumadin).
* Current use of highly protein-bound drugs including diazepam, diazoxide and lidocaine.
* Current use of digoxin.
* Any prior use of bisphosphonates, denosumab, strontium, fluoride, teriparatide or parathyroid hormone.
* Prior use of estrogen, raloxifene, calcitonin or testosterone will be allowed if discontinued more than six months previously. Low dose intra-vaginal estrogens (0.3 mg or less of conjugated equine estrogen or equivalent) may be continued throughout the study.
* Treatment with glucocorticoids in doses ≥ 5 mg prednisone daily for > 30 days in the prior year.
* Treatment with other drugs known to affect bone metabolism, e.g., anticonvulsants except benzodiazepines or gabapentin, within the prior year. Note: oral calcium supplementation, vitamin D supplementation or diuretic use that has been stable for six months are allowed).
* Treatment within the last 30 days with any drug that has not received regulatory approval.
* Metal in spine precluding spine QCT.
* Any condition that may interfere with evaluation of at least two lumbar vertebrae determined on VFA performed at time of screening. Examples include confluent aortic calcification, severe osteoarthritis, spinal fusion and lumbar spine fractures.

Ages: 60 Years to 89 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Binkley, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Osteoporosis Clinical Center and Research Program, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Daily Teriparatide (Forteo) | Monthly Cycles of Teriparatide Followed by Raloxifene
Started | 13 | 13
Completed | 12 | 13
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Daily Teriparatide (Forteo) | Monthly Cycles of Teriparatide Followed by Raloxifene | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Full Range); unit: years] | 67.7 [61.2 to 83.1] | 66.2 [56.0 to 78.8] | 67.0 [56.0 to 83.1]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 7 | 11
  >=65 years | 9 | 6 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Serum Markers of Skeletal Turnover (Serum CTX)
Description: Serum CTX was measured at all study visits following the screening visit. The outcome data is an overall average and range from all time points.
Time Frame: These were measured at the baseline and 1, 1.5, 2, 2.5, 3, 4, 5 and 6 month visits.
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | Daily Teriparatide (Forteo) | Monthly Cycles of Teriparatide Followed by Raloxifene
Number analyzed (Participants) | 13 | 13
ng/mL | 0.9887 [0.5989 to 1.4042] | 0.5445 [0.433 to 0.5838]

2. Secondary Outcome: Average Bone Mineral Density of the Spine at Baseline, 3 Months and 6 Months
Description: Spine BMD was measured at the baseline, three month and six month visits. The outcome data is an overall average and range from all time points.
Time Frame: BMD measured at the baseline, 3 month, and 6 month visits.
Measure: Mean (Full Range); unit: g/cm2
Arm/Group | Daily Teriparatide (Forteo) | Monthly Cycles of Teriparatide Followed by Raloxifene
Number analyzed (Participants) | 13 | 13
g/cm2 | 0.9599 [0.819 to 1.192] | 0.9006 [0.718 to 1.094]

3. Primary Outcome: Serum Markers of Skeletal Turnover (Serum P1NP)
Description: Serum P1NP was measured at all study visits following the screening visit. The outcome data is an overall average and range from all time points.
Time Frame: These were measured at the baseline and 1, 1.5, 2, 2.5, 3, 4, 5 and 6 month visits.
Measure: Mean (Full Range); unit: mcg/L
Arm/Group | Daily Teriparatide (Forteo) | Monthly Cycles of Teriparatide Followed by Raloxifene
Number analyzed (Participants) | 13 | 13
mcg/L | 128.7 [61.3 to 177.9] | 83.8 [52.8 to 110.8]

4. Secondary Outcome: Average Bone Mineral Density of the Proximal Femur (Hip) at Baseline, 3 Months and 6 Months
Description: Hip BMD was measured at the baseline, three month and six month visits. The outcome data is an overall average and range from all time points.
Time Frame: BMD measured at the baseline, 3 month, and 6 month visits.
Measure: Mean (Full Range); unit: g/cm2
Arm/Group | Daily Teriparatide (Forteo) | Monthly Cycles of Teriparatide Followed by Raloxifene
Number analyzed (Participants) | 13 | 13
g/cm2 | 0.7951 [0.677 to 0.939] | 0.7898 [0.667 to 0.943]

5. Secondary Outcome: Average Bone Mineral Density of the One-third Radius at Baseline, 3 Months and 6 Months
Description: One-third radius BMD was measured at the baseline, three month and six month visits. The outcome data is an overall average and range from all time points.
Time Frame: BMD measured at the baseline, 3 month, and 6 month visits.
Measure: Mean (Full Range); unit: g/cm2
Arm/Group | Daily Teriparatide (Forteo) | Monthly Cycles of Teriparatide Followed by Raloxifene
Number analyzed (Participants) | 13 | 13
g/cm2 | 0.6858 [0.6 to 0.762] | 0.687 [0.461 to 0.87]

ADVERSE EVENTS:
Arm/Group | Daily Teriparatide (Forteo) | Monthly Cycles of Teriparatide Followed by Raloxifene
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes